CLINICAL TRIAL: NCT02656160
Title: The Effect of Dalfampridine (4-aminopyridine) on Genioglossus Muscle Activity During Wakefulness and Sleep in Healthy Control Subjects
Brief Title: Effect of Dalfampridine (4-AP) on Genioglossus Muscle Activity in Healthy Adults
Acronym: APIGLOSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Andrew Wellman, Director, Sleep Disordered Breathing Lab, Brigham and Women's Hospital, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BWH-2014P001033C
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-07

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Dalfampridine (Active Comparator)
  Interventions: Drug: Dalfampridine

INTERVENTIONS:
Drug: Placebo — Placebo 3 hrs before sleep
  Arms: Placebo
Drug: Dalfampridine — Dalfampridine 10 mg extended release 3 hrs before sleep
  Arms: Dalfampridine

SUMMARY:
In this protocol the investigators will test the effect of dalfampridine (a potassium channel blocker) on genioglossus muscle activity (EMG GG) during wakefulness and sleep in healthy control subjects.

DETAILED DESCRIPTION:
Two overnight sleep studies, a placebo night and a drug night, will be performed approximately one week apart in random order. The placebo or drug will be administered 3 hours before lights out. At least 10 minutes of quiet wakefulness will be recorded to quantify the subject's awake EMG GG activity before the administration of placebo/dalfampridine.

EMG GG activity will be measured again 10 mins before lights off and during stable NREM and REM sleep (free of arousals and other artifacts).

During the second part of the night, the subjects will be connected to a modified continuous positive airway pressure (CPAP) machine (Pcrit3000, Respironics) which can provide a wide range of pressures between 20 and -20 cmH2O in order to modify upper airway pressure and measure change in EMG GG as a function of epiglottic pressure (muscle responsiveness).

ELIGIBILITY:
Inclusion Criteria:

* Healthy control subjects

Exclusion Criteria:

* Cardiovascular disease other than well controlled hypertension
* History of seizures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Disorders Research Program Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Taranto-Montemurro L, Sands SA, Azarbarzin A, Marques M, de Melo CM, Edwards BA, Eckert DJ, Messineo L, White DP, Wellman A. Effect of 4-Aminopyridine on Genioglossus Muscle Activity during Sleep in Healthy Adults. Ann Am Thorac Soc. 2017 Jul;14(7):1177-1183. doi: 10.1513/AnnalsATS.201701-006OC. PMID 28387543

RESULTS

PARTICIPANT FLOW:
Groups:
- 4-AP First, Placebo Second: 4-AP 10 mg administered 3 hours before normal sleep time on first study night, then a 1-week non-treatment period, then placebo-matching 4-AP administered 3 hours before normal sleep time on second study night.
- Placebo First, 4-AP Second: Placebo-matching 4-AP administered 3 hours before normal sleep time on first study night, then a 1-week non-treatment period, then 4-AP administered 3 hours before normal sleep time on second study night.
Period: First Study Night
Arm/Group | 4-AP First, Placebo Second | Placebo First, 4-AP Second
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0
Period: Second Study Night
Arm/Group | 4-AP First, Placebo Second | Placebo First, 4-AP Second
Started | 4 (3 subjects did not return for the second study night) | 6
Completed | 4 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Analyzed Participants: All participants who were randomized, completed both study nights, and were included in the analysis.
Arm/Group | All Analyzed Participants
Number analyzed (Participants) | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 28 [25.3 to 33.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Genioglossus Activity During Sleep Expressed as %Wakefulness Value (Before Drug/Placebo Administration).
Description: The EMG GG was quantified in arbitrary units derived from signal processing of the raw signal and as a percentage of wakefulness (%wake) for between-nights comparison of baseline sleep EMG GG activity. EMG GG analysis was performed on a breath-by-breath basis to identify a maximum value and a minimum value during inspiration and expiration, respectively (EMG GG peak and tonic). The difference between peak and tonic values was used to estimate respiratory related phasic activity. Wakefulness EMG GG values were obtained from a minimum of 10 epochs (30 s each) with the subject lying in the lateral position. Criteria for breath selection during wakefulness were (1) stable breathing (constant epiglottic pressure swings) and (2) absence of movement artifacts (i.e., swallowing, speech, yawns).
Time Frame: 1 night
Measure: Median (Inter-Quartile Range); unit: percentage of wakefulness value
Arm/Group | Placebo | Dalfampridine
Number analyzed (Participants) | 10 | 10
percentage of wakefulness value
  Tonic genioglossus activity during sleep | 166 [101 to 333] | 136 [90 to 576]
  Phasic genioglossus activity during sleep | 245 [88 to 428] | 163 [109 to 793]
Statistical Analysis 1: Comparison: Placebo vs Dalfampridine; tonic; Test type: Other; p = 0.85, Wilcoxon (Mann-Whitney) — P<0.05 considered statistically significant
Statistical Analysis 2: Comparison: Placebo vs Dalfampridine; Phasic activity; Test type: Other; p = 0.322, Wilcoxon (Mann-Whitney) — P<0.05 considered statistically significant

2. Secondary Outcome: Change in EMG GG for cmH2O Change in Epiglottic Pressure. (GG%Max/cmH2O)
Description: Effect of dalfampridine on genioglossus muscle responsiveness to increased epiglottic pressure swings during sleep in healthy controls during NREM sleep. The variation of EMG GG is expressed here as % of maximal activation.
Time Frame: 1 night
Measure: Median (Inter-Quartile Range); unit: %max/cmH2O
Arm/Group | Placebo | Dalfampridine
Number analyzed (Participants) | 10 | 10
%max/cmH2O | -0.23 [-0.57 to -0.09] | -0.36 [-1.06 to -0.1]
Statistical Analysis 1: Comparison: Placebo vs Dalfampridine; Test type: Other; p = 0.42, Wilcoxon (Mann-Whitney) — P<0.05 considered statistically significant

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Placebo | Dalfampridine
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Dalfampridine (N=10)
Headache (Nervous system disorders) | 0 (0) | 1 (1) — Headache after 1 hour from administration of dalfampridine, spontaneously recovered after approximately 1.5 hours

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes